CLINICAL TRIAL: NCT04056585
Title: Intermittent Pneumatic Compression May Reduce Brachial Plexus Block Onset Time
Brief Title: Intermittent Compression Maneuver of Upper Arm to Reduce Axillary Brachial Plexus Block Onset Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic Kwandong University (Other)
Responsible Party: Principal Investigator, Hye-Won Jeong, Assistant Professor, Catholic Kwandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CatholicKU
Record Dates: First submitted 2019-08-09; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Forearm Injuries; Hand Injuries
Keywords: brachial plexus block; intermittent pneumatic compression maneuver
MeSH Terms: conditions — Forearm Injuries; Hand Injuries

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial plexus block with intermittent pneumatic compression (Experimental): Hand and forearm surgery is performed after axillary brachial plexus block with intermittent pneumatic compression for 3 minutes.
  Interventions: Procedure: Ultrasound guided axillary plexus block; Procedure: Intermittent pneumatic compression maneuver
- Brachial plexus block (Placebo Comparator): Hand and forearm surgery is performed after axillary brachial plexus block only.
  Interventions: Procedure: Ultrasound guided axillary plexus block

INTERVENTIONS:
Procedure: Ultrasound guided axillary plexus block — Ultrasound guided axillary plexus block with 1.5% mepivacaine 30 ml
Procedure: Intermittent pneumatic compression maneuver — Following ultrasound guided axillary plexus block, the pneumatic compression maneuver of upper arm is composed of 6 repeated inflation-deflation periods; inflation with a pressure of 200 mmHg for 30 seconds and deflation for 10 seconds each.
  Arms: Brachial plexus block with intermittent pneumatic compression

SUMMARY:
This study evaluates the addition of intermittent pneumatic compression maneuver to axillary brachial plexus block in forearm and hand surgery. Half of participants will receive axillary brachial plexus block and intermittent pneumatic compression maneuver, while the other half will receive only axillary brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

1. adults between ages of 20 and 50
2. patients who are scheduled forearm and hand surgery with axillary brachial plexus block
3. American Society of Anesthesiologists Physical Status classification 1 or 2
4. patients who voluntarily agree to participate in the trial

Exclusion Criteria:

1. patients who are pregnant or lactating
2. patient who does not agree to participate in the study
3. patient with side effects on local anesthetics
4. patient with neurologic deficit of upper arm
5. patients with comorbidities of cardiac, pulmonary, renal, cerebral, and hepatic systems
6. patients with peripheral vascular disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Time to achieve complete sensory block | 1 hour
  Defined as the time to reach an absent sensation in the pinprick test at all four nerve distributions (ulnar nerve, radial nerve, median nerve, and musculocutaneous nerve)

SECONDARY OUTCOMES:
Time to achieve surgical anaesthesia | 1 hour
  Defined as the time to reach an absent sensation in the pinprick test and reduced power at all four nerve distributions (ulnar nerve, radial nerve, median nerve, and musculocutaneous nerve)

CONTACTS AND LOCATIONS:
Locations (1):
- International St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No